CLINICAL TRIAL: NCT06311864
Title: Real-World Observational Study on Patient-Reported Outcomes in the Treatment of Insomnia with Daridorexant in Canada
Status: Enrolling by invitation | Type: Observational
Sponsor: PeriPharm (Other)
Collaborators: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Principal Investigator, Jean Lachaine, Principal Investigator, PeriPharm
Other Study IDs: PROxy240215
Record Dates: First submitted 2024-03-06; First posted 2024-03-15 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Insomnia
Keywords: daridorexant; dual orexin receptor antagonist; real-world; observational; quality of life; work productivity; insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — daridorexant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- daridorexant: Patients who have been newly prescribed oral tablets of daridorexant 50 mg to treat their insomnia
  Interventions: Drug: Daridorexant 50 mg

INTERVENTIONS:
Drug: Daridorexant 50 mg — As indicated by the physician
  Other Names: QUVIVIQ

SUMMARY:
The purpose of this observational study is to evaluate the impact of daridorexant on quality of life, work productivity and insomnia symptoms in Canadian adults suffering from insomnia.

DETAILED DESCRIPTION:
Participating physicians will identify potential participants based on their medical judgment for a new prescription of QUVIVIQ® (daridorexant) 50 mg. Physicians will discuss with the potential participant in person to briefly describe the study (purpose, confidentiality, questionnaires, as well as compensation). Potential participants interested in participating in the study will be asked to give their authorization to share with the PROxy Network their contact information by signing an authorization form. A designated PROxy team member will then contact the potential participant to explain the study in more details and to assess the eligibility. If the potential participant agrees to participate and provides verbal consent, he/she will be invited to visit the Participant Portal on the PROxy website to sign the ICF and complete the online baseline questionnaires.

Five days prior to each study timepoint (1 month, 2 months and 3 months following baseline questionnaire completion), participants will receive an email inviting them to fill their study questionnaires. This e-mail will be sent every other day to the participant who have not completed the questionnaires. In the case where a participant has not completed the questionnaires within a period of 5 days after the first email was sent, a call will be made by a designated PROxy team member to remind the patient to complete the questionnaire. Participants who don't complete the questionnaires in the 5 days following the call will be excluded from this timepoint analysis.

ELIGIBILITY:
Inclusion Criteria:

* Signed ICF prior to any study-mandated procedure.
* Has received a first prescription of daridorexant 50 mg to treat insomnia, treatment start has not exceeded 7 days prior to enrollment.
* Ability to read and understand French or English.

Exclusion Criteria:

* Patients participating in a clinical trial.
* History of daridorexant use in the past (i.e., samples provided by the physician before prescription).
* Taking a concomitant medication to treat insomnia.
* Already started daridorexant more than 7 days prior to enrollment.The 7-day period is necessary to allow flexibility between the time of prescription and PROxy first contact to participant. Beyond this 7-day period, patients may already have experienced benefits from daridorexant. To minimize bias in baseline results, these patients will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients identified by 10 participating physicians in 4 provinces across Canada (Quebec, Ontario, Alberta, British Columbia)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Quality of Life | Month 1, Month 2, Month 3
  QoL will be measured using the SF-36 questionnaire, a self-administered and validated questionnaire. The percentage change from baseline in each domain of the SF-36 will be assessed at Month 1, Month 2 and Month 3.
Change from Baseline in Work Productivity Loss | Month 1, Month 2, Month 3
  Work productivity loss will be measured using the Work Productivity and Activity Impairment for Specific Health Problem (WPAI:SHP), a self-administered and validated 6-item questionnaire designed to assess the impact of a health condition on work productivity and daily activities for a specific disease/condition (in this case, insomnia). The percentage change from baseline on the WPAI:SHP score at month 1, month 2 and month 3 will be assessed.
Change from Baseline in the Severity of Insomnia Symptoms | Month 1, Month 2, Month 3
  Severity of insomnia symptoms will be measured using the Insomnia Severity Index (ISI) questionnaire, a self-administered, validated, 7-item questionnaire, designed to assess the severity of insomnia symptoms. The ISI will be assessed at Month 1, Month 2, and Month 3.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Lachaine, PhD, Principal Investigator — PeriPharm
Locations (1):
- PROxy Network, an initiative of PeriPharm inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No